CLINICAL TRIAL: NCT01421706
Title: Effects of Clopidogrel and Clarithromycin on the Disposition of Sibutramine and Its Active Metabolites M1 and M2 in Relation to CYP2B6*6 Polymorphism
Brief Title: Effects of Clopidogrel and Clarithromycin on the Oral Disposition of Sibutramine in Healthy Subjects
Acronym: sibu
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Inje University (Other)
Responsible Party: Principal Investigator, Jae-Gook Shin, Professor, Inje University
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: 08-073
Record Dates: First submitted 2011-08-22; First posted 2011-08-23 (Estimated); Last update posted 2012-09-18 (Estimated); Status verified 2012-09

CONDITIONS: Healthy
Keywords: clarithromycin; sibutramine; clopidogrel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- sibutramine-clopidogrel (Active Comparator): sibutramine-clopidogrel
  Interventions: Drug: Sibutramine-clopidogrel
- sibutramine-clarithromycin (Active Comparator): sibutramine-clarithromycin
  Interventions: Drug: sibutramine-Clarithromycin

INTERVENTIONS:
Drug: Sibutramine-clopidogrel — Sibutramine-clopidogrel
  Arms: sibutramine-clopidogrel
Drug: sibutramine-Clarithromycin — sibutramine-Clarithromycin
  Arms: sibutramine-clarithromycin

SUMMARY:
Effects of clopidogrel and clarithromycin on the oral disposition of sibutramine in healthy subjects

DETAILED DESCRIPTION:
1. Plasma concentrations of sibutramine and its two active metabolites after single oral dose of sibutramine were determined in Korean healthy male subjects with different CYP2B6 genotypes (CYP2B6*1/*1, *1/*6 and *6/*6), either alone or after four-day pretreatment with clopidogrel or clarithromycin.

ELIGIBILITY:
Inclusion Criteria:

* must be healthy volunteer

Exclusion Criteria:

* must not be under 18 years old

Ages: 19 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2008-07; Primary Completion 2009-07 (Actual); Study Completion 2009-07 (Actual)

PRIMARY OUTCOMES:
effects of clopidogrel and clarithromycin on the disposition of sibutramine | one year
  the effects of clopidogrel and clarithromycin on the disposition of sibutramine and its two active metabolites M1 and M2 in vivo in relation to CYP2B6*6 genetic polymorphism have been evaluated in Korean healthy subjects.

CONTACTS AND LOCATIONS:
Overall Officials: JaeGook Shin, MD,PhD, Principal Investigator — Inje University